CLINICAL TRIAL: NCT06352645
Title: Evaluation of Safety and Efficacy of Bixdo Ultra Compact Water Flosser in Addition to Toothbrushing-A 8-week Randomized Controlled Trial
Brief Title: Evaluation of Safety and Efficacy of Bixdo Ultra Compact Water Flosser
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tufts University (Other)
Collaborators: Guang Dong Bixdo Health Technology Co.,Ltd (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00004879
Record Dates: First submitted 2024-04-02; First posted 2024-04-08 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Plaque Induced Gingivitis

STUDY DESIGN:
Intervention Model Description: randomized controlled clinical trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Interventional Group (Experimental): Those randomized into the interventional group will be asked to use the Bixdo Ultra Compact Water Flosser twice a day for 8 weeks.
  Interventions: Device: Bixdo Ultra Compact Water Flosser
- Control Group (Active Comparator): Those randomized into the control group will be asked to only use the study provided manual toothbrush and toothpaste twice a day for 8 weeks.
  Interventions: Device: Manual toothbrush

INTERVENTIONS:
Device: Bixdo Ultra Compact Water Flosser — Use of water flosser, in addition to standard tooth brushing, twice a day for 8 weeks.
  Arms: Interventional Group
Device: Manual toothbrush — For those in the control group, they will be asked to use only the study-provided manual toothbrush, twice a day for 8 weeks.
  Arms: Control Group

SUMMARY:
The objective of the present randomized controlled trial is to evaluate the safety and efficacy of the use of Bixdo A30 Pro Ultra Compact Water Flosser (also referred to as the "Bixdo A30 Portable Water Flosser Travel Set") in addition to a manual toothbrush on clinical parameters of inflammation and bacterial plaque removal.

ELIGIBILITY:
Inclusion Criteria:

1. Participants between the age of 18 - 70 years old.
2. Having at least 20 natural teeth in their dentition - excluding third molars.
3. In good overall systemic health, in the opinion of the investigator.
4. In good dental health with no visible carious lesions, periodontitis, orthodontic appliances, or removable partial dentures.
5. No hard or soft tissue lesions.
6. Subjects with moderate or severe plaque-induced gingivitis: a minimum of 50% BOP, 1.75 modified gingival index (MGI), and 0.60 Rustogi Modification of the Navy Plaque Index (RMNPI) and PPD ≤5 mm.
7. Subjects who agree to delay dental prophylaxis, elective dental treatment, and cosmetic procedures (i.e. tooth whitening, crowns) for the duration of the study
8. For the main study only: Subjects who agree to refrain from using any non-study dental device or oral care products for the duration of the study, return for scheduled visits, and comply with all study procedures.

Exclusion Criteria:

1. Systemic disease self-reported that has an impact on periodontal status (e.g., diabetes mellitus, HIV/AIDS, rheumatoid arthritis).
2. History of any autoimmune disease (e.g., pSS, SLE, psoriasis, IBS).
3. History of immunosuppressive chemotherapy or history of any disease known to severely compromise immune function (e.g., cytomegalovirus infection) within the last 5 years.
4. Any acute intraoral infection (e.g., herpetic gingivostomatitis, herpangina, abscesses).
5. Patients with visible carious lesions, periodontitis, orthodontic appliances, or removable partial dentures.
6. Patients with mild plaque-induced gingivitis: < 50% BOP, <1.75 modified gingival index (MGI), and <0.60 Rustogi Modification of the Navy Plaque Index (RMNPI) and PPD ≤5 mm.
7. Patients with PPD >5 mm.
8. Need for antibiotic premedication for routine dental procedures.
9. Use of antibiotics within the last 3 months.
10. Daily use of steroids or non-steroid anti-inflammatory therapy within the last 3-months.
11. Patients who self-report pregnancy or lactation (hormonal changes that can affect periodontal health and aggravate existing periodontal disease).
12. Current smokers.
13. Inability or unwillingness to sign informed consent form.
14. Patients who do not agree to delay dental prophylaxis, elective dental treatment, and cosmetic procedures (i.e. tooth whitening, crowns).
15. For the main study only: Patients who do not agree to refrain from using any non-study dental device or oral care products, return for scheduled visits, and comply with all study procedures.
16. Anything that would place the individual at increased risk or preclude the individual's full compliance with or completion of the study at the discretion of the investigators.
17. For the main study only: Patients who need assistance from others to perform their daily oral hygiene practices or read the manual of instructions that come with the at-home product.
18. Those not fluent in English

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 165 (Estimated)
Dates: Start 2025-03-04 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Inflammation Reduction | 8 weeks
  At each of the three study visits, the examiners will conduct a periodontal clinical exam, following standard of care procedure, to evaluate the levels of inflammation in the gingiva of subjects in both the intervention and control groups.
Bacterial plaque removal | 8 weeks
  At each of the three study visits, subjects will be given dental plaque erythrosine disclosing agents (Sunstar GUM® RED-COTE®) to assess the level of plaque on the subjects teeth

CONTACTS AND LOCATIONS:
Overall Officials: Mabi Singh, Principal Investigator — Tufts University School of Dental Medicine
Locations (1):
- Tufts University School of Dental Medicine, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] GBD 2017 Disease and Injury Incidence and Prevalence Collaborators. Global, regional, and national incidence, prevalence, and years lived with disability for 354 diseases and injuries for 195 countries and territories, 1990-2017: a systematic analysis for the Global Burden of Disease Study 2017. Lancet. 2018 Nov 10;392(10159):1789-1858. doi: 10.1016/S0140-6736(18)32279-7. Epub 2018 Nov 8. PMID 30496104
- [Background] Tonetti MS, Claffey N; European Workshop in Periodontology group C. Advances in the progression of periodontitis and proposal of definitions of a periodontitis case and disease progression for use in risk factor research. Group C consensus report of the 5th European Workshop in Periodontology. J Clin Periodontol. 2005;32 Suppl 6:210-3. doi: 10.1111/j.1600-051X.2005.00822.x. No abstract available. PMID 16128839
- [Background] Bashir NZ. Update on the prevalence of untreated caries in the US adult population, 2017-2020. J Am Dent Assoc. 2022 Apr;153(4):300-308. doi: 10.1016/j.adaj.2021.09.004. Epub 2021 Dec 22. PMID 34952680
- [Background] Tarnow DP. Increasing Prevalence of Peri-implantitis: How Will We Manage? J Dent Res. 2016 Jan;95(1):7-8. doi: 10.1177/0022034515616557. No abstract available. PMID 26701918
- [Background] Kassebaum NJ, Bernabe E, Dahiya M, Bhandari B, Murray CJ, Marcenes W. Global burden of severe periodontitis in 1990-2010: a systematic review and meta-regression. J Dent Res. 2014 Nov;93(11):1045-53. doi: 10.1177/0022034514552491. Epub 2014 Sep 26. PMID 25261053
- [Background] Eke PI, Borgnakke WS, Genco RJ. Recent epidemiologic trends in periodontitis in the USA. Periodontol 2000. 2020 Feb;82(1):257-267. doi: 10.1111/prd.12323. PMID 31850640
- [Background] Cochran DL. Inflammation and bone loss in periodontal disease. J Periodontol. 2008 Aug;79(8 Suppl):1569-76. doi: 10.1902/jop.2008.080233. PMID 18673012
- [Background] Kinane DF, Stathopoulou PG, Papapanou PN. Periodontal diseases. Nat Rev Dis Primers. 2017 Jun 22;3:17038. doi: 10.1038/nrdp.2017.38. PMID 28805207
- [Background] Linden GJ, Herzberg MC; Working group 4 of joint EFP/AAP workshop. Periodontitis and systemic diseases: a record of discussions of working group 4 of the Joint EFP/AAP Workshop on Periodontitis and Systemic Diseases. J Clin Periodontol. 2013 Apr;40 Suppl 14:S20-3. doi: 10.1111/jcpe.12091. PMID 23627330
- [Background] Genco RJ, Van Dyke TE. Prevention: Reducing the risk of CVD in patients with periodontitis. Nat Rev Cardiol. 2010 Sep;7(9):479-80. doi: 10.1038/nrcardio.2010.120. PMID 20725103
- [Background] Lalla E, Papapanou PN. Diabetes mellitus and periodontitis: a tale of two common interrelated diseases. Nat Rev Endocrinol. 2011 Jun 28;7(12):738-48. doi: 10.1038/nrendo.2011.106. PMID 21709707
- [Background] Lundberg K, Wegner N, Yucel-Lindberg T, Venables PJ. Periodontitis in RA-the citrullinated enolase connection. Nat Rev Rheumatol. 2010 Dec;6(12):727-30. doi: 10.1038/nrrheum.2010.139. Epub 2010 Sep 7. PMID 20820197
- [Background] Whitmore SE, Lamont RJ. Oral bacteria and cancer. PLoS Pathog. 2014 Mar 27;10(3):e1003933. doi: 10.1371/journal.ppat.1003933. eCollection 2014 Mar. No abstract available. PMID 24676390
- [Background] Madianos PN, Bobetsis YA, Offenbacher S. Adverse pregnancy outcomes (APOs) and periodontal disease: pathogenic mechanisms. J Clin Periodontol. 2013 Apr;40 Suppl 14:S170-80. doi: 10.1111/jcpe.12082. PMID 23627327
- [Background] Heitz-Mayfield LJ, Trombelli L, Heitz F, Needleman I, Moles D. A systematic review of the effect of surgical debridement vs non-surgical debridement for the treatment of chronic periodontitis. J Clin Periodontol. 2002;29 Suppl 3:92-102; discussion 160-2. doi: 10.1034/j.1600-051x.29.s3.5.x. PMID 12787211
- [Background] Chapple IL, Van der Weijden F, Doerfer C, Herrera D, Shapira L, Polak D, Madianos P, Louropoulou A, Machtei E, Donos N, Greenwell H, Van Winkelhoff AJ, Eren Kuru B, Arweiler N, Teughels W, Aimetti M, Molina A, Montero E, Graziani F. Primary prevention of periodontitis: managing gingivitis. J Clin Periodontol. 2015 Apr;42 Suppl 16:S71-6. doi: 10.1111/jcpe.12366. PMID 25639826
- [Background] Edlund P, Bertl K, Pandis N, Stavropoulos A. Efficacy of power-driven interdental cleaning tools: A systematic review and meta-analysis. Clin Exp Dent Res. 2023 Feb;9(1):3-16. doi: 10.1002/cre2.691. Epub 2022 Dec 23. PMID 36562267
- [Background] Xu X, Zhou Y, Liu C, Zhao L, Zhang L, Li H, Li Y, Cheng X. Effects of water flossing on gingival inflammation and supragingival plaque microbiota: a 12-week randomized controlled trial. Clin Oral Investig. 2023 Aug;27(8):4567-4577. doi: 10.1007/s00784-023-05081-4. Epub 2023 May 25. PMID 37231271
- [Background] Lyle DM, Qaqish JG, Goyal CR, Schuller R. Efficacy of the Use of a Water Flosser in Addition to an Electric Toothbrush on Clinical Signs of Inflammation: 4-Week Randomized Controlled Trial. Compend Contin Educ Dent. 2020 Mar 1;41(3):170-177. Epub 2020 Jan 1. PMID 31904246
- [Background] Slot DE, Valkenburg C, Van der Weijden GAF. Mechanical plaque removal of periodontal maintenance patients: A systematic review and network meta-analysis. J Clin Periodontol. 2020 Jul;47 Suppl 22:107-124. doi: 10.1111/jcpe.13275. PMID 32716118
- [Background] Tyler D, Kang J, Goh HH. Effectiveness of Waterpik(R) for oral hygiene maintenance in orthodontic fixed appliance patients: A randomised controlled trial. J Orthod. 2023 Dec;50(4):367-377. doi: 10.1177/14653125231173708. Epub 2023 May 19. PMID 37203873
- [Background] Sawan N, Ben Gassem A, Alkhayyal F, Albakri A, Al-Muhareb N, Alsagob E. Effectiveness of Super Floss and Water Flosser in Plaque Removal for Patients Undergoing Orthodontic Treatment: A Randomized Controlled Trial. Int J Dent. 2022 Aug 31;2022:1344258. doi: 10.1155/2022/1344258. eCollection 2022. PMID 36090126
- [Background] Lobene RR, Weatherford T, Ross NM, Lamm RA, Menaker L. A modified gingival index for use in clinical trials. Clin Prev Dent. 1986 Jan-Feb;8(1):3-6. No abstract available. PMID 3485495
- [Background] Rustogi KN, Curtis JP, Volpe AR, Kemp JH, McCool JJ, Korn LR. Refinement of the Modified Navy Plaque Index to increase plaque scoring efficiency in gumline and interproximal tooth areas. J Clin Dent. 1992;3(Suppl C):C9-12. PMID 1306676
- [Background] Goyal CR, Lyle DM, Qaqish JG, Schuller R. The addition of a water flosser to power tooth brushing: effect on bleeding, gingivitis, and plaque. J Clin Dent. 2012;23(2):57-63. PMID 22779218
- See also: Adverse Event Reporting to IRBs - Improving Human Subject Protection — https://www.fda.gov/regulatory-information/search-fda-guidance-documents/adverse-event-reporting-irbs-improving-human-subject-protection